CLINICAL TRIAL: NCT00509002
Title: Phase II Study of ZD1839 (Iressa®), Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor in Patients With Advanced, Recurrent or Metastatic Salivary Gland Cancer (IRUSIRES0198)
Brief Title: Iressa Study in Patients With Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0089; NCI-2010-00744 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Salivary Gland Cancer
Keywords: Salivary Gland Cancer; Iressa; ZD1839
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adenoid Cystic Salivary Gland Carcinoma Group (Experimental): Participants receive Gefitinib daily by mouth until progressive disease, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Gefitinib
- Other Carcinoma of Salivary Gland Group (Experimental): Participants receive Gefitinib daily by mouth until progressive disease, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg by mouth once a day, every day, at about same time in morning.
  Other Names: Iressa; ZD1839

SUMMARY:
The goal of this clinical research study is to learn if ZD1839 (Iressa®, gefitinib can help to shrink or slow the growth of advanced, recurrent, or metastatic salivary gland cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Epidermal growth factor receptor (EGFR) may be involved in certain types of cancer, including squamous cell carcinoma of the skin. When EGFR is stimulated, a series of chemical reactions starts that results in a tumor being "told" to grow. ZD1839 (Iressa® or Gefitinib) tries to stop these reactions by blocking EGFR. This may stop tumors from growing.

If you are eligible to take part in this study, you will take gefitinib treatment by mouth once a day, every day, at about the same time in the morning. It can be taken with or without food. If you forget to take a dose, the last missed dose should be taken as soon as you remember, as long as it is at least 12 hours before the next dose is due to be taken.

Every four weeks during treatment, you will have a physical exam and blood (around 3-4 teaspoons) will be collected for routine tests. If you have skin lesions, the lesions will be measured and photographed for research purposes. You cannot be identified from the pictures. You will also be asked about any side effects you may be experiencing. If your doctor feels it is necessary, you may have more frequent check-ups.

Every eight weeks during treatment, you will have imaging tests. The imaging tests include, a chest x-ray and a CT scan or MRI of the head and neck area. You may also have CT scans of other areas of the body. These tests are being done to check on the status of the disease.

You will continue to take gefitinib as long as the disease is responding to treatment. If at any time during the study the disease becomes worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Sometimes, new information becomes available that may influence your decision to continue in the study. The following new information is available:

Results from two large studies showed that there was no benefit from adding gefitinib to chemotherapy with platinum and one other chemotherapy drug when given as the first treatment for non-small cell lung cancer (NSCLC). Therefore, gefitinib is not approved for use in combination with chemotherapy in the treatment of NSCLC.

This is an investigational study. The FDA has authorized gefitinib for use in cancer research. Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed salivary gland carcinoma.
2. Patients with advanced or recurrent salivary gland cancer who are not candidates for curative surgery or radiotherapy.
3. Measurable disease per the RECIST criteria. For disease occurring in previously irradiated field, there must be confirmed progression prior to the date registration and more than three months after completion of radiotherapy
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Prior central nervous system (CNS) involvement by tumor is permissible if previously treated and clinically stable for two weeks after completion of treatment.
6. At least a 2-week recovery from prior therapy toxicity.
7. Provision of written informed consent.
8. Childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (IUD, birth control pills, or barrier device) during and for 3 months after completion of trial therapy.

Exclusion Criteria:

1. Known severe hypersensitivity to or any of the excipients of this product.
2. Other coexisting malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma, squamous cell carcinoma of the skin, or cervical cancer in situ.
3. Concomitant use of phenytoin, carbamazepine, rifampicin, phenobarbital, or St John's Wort or CYP3A4 (e.g. itraconazole, ketoconazole)
4. Treatment with a investigational drug within 28 days before Day 1 of trial treatment.
5. Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy (except alopecia)
6. Incomplete healing from previous surgery.
7. Serum creatinine level greater than CTC grade 2.
8. Women who are pregnant or breast feeding.
9. Prior or other EGFR inhibiting agents.
10. Serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR).
11. Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
12. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases or greater than 5 times the ULRR in the presence of liver metastases.
13. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial.
14. Uncontrolled seizure disorder, active neurological disease, or greater than Grade 2 neuropathy.
15. Keratoconjunctivitis sicca or incompletely treated eye infection.
16. Abnormal marrow function as defined as absolute neutrophil count <1,500/ul or platelets <100,000/ul.
17. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 3 years previously with no evidence of recurrence; prior low grade [Gleason score less than 6] localized prostate cancer is allowed).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Blumenschein, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jakob JA, Kies MS, Glisson BS, Kupferman ME, Liu DD, Lee JJ, El-Naggar AK, Gonzalez-Angulo AM, Blumenschein GR Jr. Phase II study of gefitinib in patients with advanced salivary gland cancers. Head Neck. 2015 May;37(5):644-9. doi: 10.1002/hed.23647. Epub 2015 Mar 30. PMID 24585506
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2004 to October 2006. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Gefitinib: Gefitinib 250 mg daily by mouth until progressive disease, unacceptable toxicity or patient withdrawal.
Period: Overall Study
Arm/Group | Gefitinib
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of ZD1839 in Patients With Advanced or Recurrent Salivary Gland Cancer Who Are Not Candidate for Curative Surgery or Radiotherapy
Description: The modified Response Evaluation Criteria in Solid tumors (RECIST) criteria was used for objective tumor response assessment. Complete Response (CR): Disappearance all target lesions; Partial Response (PR): >30% decrease in sum longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): >20% increase in sum LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of one or > new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started. Response rate estimated by Gehan's Phase II clinical trial design.
Time Frame: Every 4 weeks until progressive disease, unacceptable toxicity or patient withdrawal
Measure: Count of Participants; unit: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 37
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 18
  Progressive Disease | 13
  Inevaluable | 6

ADVERSE EVENTS:
Time Frame: Adverse events collected every four weeks during treatment at regular assessment, participation expected up to 12 months.
Arm/Group | Gefitinib
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 37/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib (N=37)
Anorexia (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 30 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8)
Fatigue (General disorders) | 15 (16)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes